CLINICAL TRIAL: NCT07395219
Title: Prospective Evaluation of the Safety and Efficacy of Transoral Incisionless Fundoplication 2.0 in the Management of Reflux: a European Registry
Brief Title: European TIF2.0 Registry
Acronym: EURO-TIF
Status: Enrolling by invitation | Type: Observational
Sponsor: Cleveland Clinic London (Other)
Responsible Party: Sponsor
Other Study IDs: CCL-2021-TIF
Record Dates: First submitted 2025-11-25; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Gastro -Oesophagal Reflux; Laryngo-pharyngeal Reflux
Keywords: TIF; cTIF; GORD; GERD; Endoscopic intervention; Endoscopy; reflux
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Patients with gastro-oesophageal reflux disease or laryngo-pharyngeal reflux
  Interventions: Device: Transoral incisionless fundoplication with or without concomitant hiatal hernia repair with the EsophyX device

INTERVENTIONS:
Device: Transoral incisionless fundoplication with or without concomitant hiatal hernia repair with the EsophyX device — Transoral Incisionless Fundoplication (TIF):
  The TIF procedure is an endoscopic, minimally invasive intervention designed to reconstruct the gastro-oesophageal valve and restore its function as a reflux barrier, without external incisions. The procedure is performed transorally using the EsophyX device under general anaesthesia. The device enables the creation of a 270° to 300° esophagogastric fundoplication.
  Concomitant TIF (cTIF):
  The cTIF procedure combines a laparoscopic hiatal hernia repair with the TIF performed in the same session. Patients with a hiatal hernia greater than 2 cm undergo laparoscopic reduction and crural repair, followed immediately by the TIF procedure using the EsophyX device. This combined approach addresses both the anatomical defect of the hiatal hernia and the functional deficiency of the gastro-oesophageal valve.
  Other Names: TIF; cTIF

SUMMARY:
This is a European, multi-centre, prospective registry that aims to determine the safety and efficacy of transoral incisionless fundoplication, with or without concomitant hiatal hernia repair, for the treatment of patients with gastro-oesophageal reflux disease (GORD).

ELIGIBILITY:
Inclusion Criteria:

* Any adult patient (≥18 years old) undergoing TIF2.0 or cTIF, at a participating centre, who can understand and sign the informed consent form, and is conducted in line with local institutional review board approval and recommendations.

Exclusion Criteria:

* There are no specific exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with gastro-oesophageal reflux disease or laryngo-pharyngeal reflux undergoing transoral incisionless fundoplication with or without concomitant hiatal hernia repair
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-08-01 (Estimated)

PRIMARY OUTCOMES:
Gastroesophageal reflux disease health-related quality of life questionnaire (GERD-HRQL) | 6-months, 1-year, 2-year, 3-years, 5-, years
  Change in reflux-specific quality of life questionnaires
  (The GERD-HRQL used in the study is composed of 16 questions related to symptoms of heartburn, regurgitation, swallowing and overall satisfaction. Each question provides a scaled score between 0-5 (0=no symptoms, 5= Symptoms incapacitating to do daily activities) with a total score of 75.)
Reflux symptom index (RSI) | 6-months, 1-year, 2-years, 3-years, 5-years
  Change in reflux-specific quality of life questionnaire
  (The RSI used in the study is composed of 9 questions related to atypical symptoms of reflux or 'LPR'. Each question provides a scaled score between 0-5 (0=no problems, 5=severe problems) with a total score of 45.)
Proton pump inhibitor and/or histamine-2 receptor antagonist use | 6-months, 1-year, 2-years, 3-years, 5-years
  Change in acid suppression use

SECONDARY OUTCOMES:
Physiological reflux testing | up to 5-years
  Change in pH physiological testing
Procedural outcomes (technical success) | 30-days
  Defined as successful completion of all steps of the cTIF or TIF2.0 procedure in the same sitting
Procedural outcomes (duration) | 30-days
  Total length of the procedure in minutes
Procedural outcomes (length of hospital stay | 30-days
  The time in days from procedure to discharge from hospital
Adverse events | up to 30-days
  Adverse events (AE) following TIF2.0 according to the AGREE classification
Adverse events of special interest | Up to 5-years
  Subjective reporting of dysphagia, excessive belching or inability to belch, significant bloating and/or distension, and persistent nausea and vomiting.
Need for revisional procedure | Up to 5-years
  The need for repreat endoscopic or surgical intervention due to recurrence of symptoms, failure of procedure of adverse events

CONTACTS AND LOCATIONS:
Locations (7):
- Department of General Surgery, Medical University of Vienna, Vienna, Austria
- Gemelli Isola, Rome, Italy
- University Hospital for Digestive Surgery, Belgrade, Serbia
- Intesto, Bern, Switzerland
- Memorial bahçelievler hospital, Istanbul, Turkey (Türkiye)
- Cleveland Clinic, Abu Dhabi, United Arab Emirates
- Cleveland Clinic London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared publicly. Data will be available only to investigators at participating study centers for the purpose of study coordination, monitoring, and analysis in accordance with the study protocol and applicable data protection regulations. Broader sharing of IPD is not planned due to confidentiality considerations and data use agreements established with participating institutions.

REFERENCES:
- [Background] Testoni S, Hassan C, Mazzoleni G, Antonelli G, Fanti L, Passaretti S, Correale L, Cavestro GM, Testoni PA. Long-term outcomes of transoral incisionless fundoplication for gastro-esophageal reflux disease: systematic-review and meta-analysis. Endosc Int Open. 2021 Feb;9(2):E239-E246. doi: 10.1055/a-1322-2209. Epub 2021 Feb 3. PMID 33553587
- [Background] Demartini B, Nistico V, D'Agostino A, Priori A, Gambini O. Early Psychiatric Impact of COVID-19 Pandemic on the General Population and Healthcare Workers in Italy: A Preliminary Study. Front Psychiatry. 2020 Dec 22;11:561345. doi: 10.3389/fpsyt.2020.561345. eCollection 2020. PMID 33414728
- [Background] Cristol DA, Evers DC. The impact of mercury on North American songbirds: effects, trends, and predictive factors. Ecotoxicology. 2020 Oct;29(8):1107-1116. doi: 10.1007/s10646-020-02280-7. Epub 2020 Sep 24. PMID 32970279
- [Background] Rahimi Z, Ghorbani-Shahna F, Bahrami A. Design, Implementation, and Evaluation of Industrial Ventilation Systems and Filtration for Silica Dust Emissions from a Mineral Processing Company. Indian J Occup Environ Med. 2021 Oct-Dec;25(4):192-197. doi: 10.4103/ijoem.IJOEM_55_19. Epub 2021 Dec 31. PMID 35197669
- [Background] Globig P, Willumeit-Romer R, Martini F, Mazzoni E, Luthringer-Feyerabend BJC. Slow degrading Mg-based materials induce tumor cell dormancy on an osteosarcoma-fibroblast coculture model. Bioact Mater. 2021 Dec 30;16:320-333. doi: 10.1016/j.bioactmat.2021.12.031. eCollection 2022 Oct. PMID 35386318
- [Background] Jaruvongvanich VK, Matar R, Reisenauer J, Janu P, Mavrelis P, Ihde G, Murray M, Singh S, Kolb J, Nguyen NT, Thosani N, Wilson EB, Zarnegar R, Chang K, Canto MI, Abu Dayyeh BK. Hiatal hernia repair with transoral incisionless fundoplication versus Nissen fundoplication for gastroesophageal reflux disease: A retrospective study. Endosc Int Open. 2023 Jan 4;11(1):E11-E18. doi: 10.1055/a-1972-9190. eCollection 2023 Jan. PMID 36618876
- [Background] Mattei C, Tricoire-Leignel H, Legros C, Lewis RJ, Molgo J. Editorial: Pharmacological Aspects of Ligand-Gated Ion Channels as Targets of Natural and Synthetic Agents. Front Neurosci. 2022 Apr 8;16:895299. doi: 10.3389/fnins.2022.895299. eCollection 2022. No abstract available. PMID 35464319